CLINICAL TRIAL: NCT05783167
Title: Self-collected Cervical Cancer Screening Samples for Detection of Human Papillomavirus in HIV-positive Women - a Pilot Study of Self-collected Vaginal and Urine Samples
Brief Title: Self-collected Vaginal and Urine Samples in HIV-positive Women
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Universiteit Antwerpen (Other); Randers Regional Hospital (Other); Bandim Health Project (Other)
Responsible Party: Sponsor
Other Study IDs: R351-A20092
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-03

CONDITIONS: HIV Infections; HPV-Related Cervical Carcinoma; Cervical Cancer; Coinfection, HIV
Keywords: Cervical cancer screening; Self-sampling; Urine sample; Vaginal sample
MeSH Terms: conditions — HIV Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HIV-positive females in Guinea-Bissau: The study is conducted on female HIV-infected patients in the Nationwide HIV-cohort at the 9 biggest HIV-clinics in Guinea-Bissau.
  Participants will be invited to enroll in the project when they present to the HIV-clinics for HIV-treatment and consultations.
  Interventions: Diagnostic Test: Self-sampling for HPV infection

INTERVENTIONS:
Diagnostic Test: Self-sampling for HPV infection — After informed consent has been provided, the woman will be asked to collect firstly a first-void urine sample using the Collipee device and secondly to collect a vaginal self-sample using the dry Evalyn® Brush device. Socioeconomic, demographic and clinical data will be collected in the Bissau HIV Cohort database and through study questionnaires to collect background information on risk factors for HPV persistence and development of cervical cancer (HIV genotype, immune status, parity). Questionnaires will collect additional information on the acceptance of cervical screening measures to better evaluate the feasibility of implementing self-collected screening among HIV infected women in Guinea-Bissau.
  Other Names: Collipee; Evalyn Brush

SUMMARY:
This study assesses topics as Human Immunodeficiency Virus (HIV), Human Papilloma Virus (HPV), and cancer screening methods. The focus will be on evaluating feasibility of implementing novel cancer screening modalities in a low-resource setting in Guinea-Bissau and further to estimate the prevalence of the precancerous virus HPV amongst women living with HIV. In the study the investigators will collect urinary and vaginal self-samples for HPV testing, and further evaluate the feasibility of implementing the devices as screening modalities through questionnaires given to the women.

DETAILED DESCRIPTION:
This pilot study will partly take place at the outpatient HIV clinic, based in the Hospital National Simão Mendes (HNSM) in the capital city Bissau, Guinea-Bissau. HNSM is the main hospital in Bissau, and the HIV clinic is the biggest HIV treatment center in Guinea-Bissau in terms of patients on follow-up. The Bissau Nationwide HIV Cohort is a clinical HIV Cohort started in 2007. As of today, the investigators collect data from 9 outpatient HIV clinics in the country, and samples will be collected from all 9 clinics.

Study participants who present at the HIV clinic will be thoroughly instructed in correct usage of the vaginal and urine devices by trained healthcare workers. At the HIV clinics, facilities will be available for the women to conduct self-sampling in privacy, before handing in the samples. At the local laboratory, the dry brush head will be suspended in Thinprep medium and stored until shipment to Denmark. The urine samples will be stored at room temperature for up to 7 days before transferred to a -20º freezer until shipment to Denmark.

Analyses: vaginal and urine samples will be analyzed at Randers Regional Hospital using the Cobas 4800 HPV DNA test. The Department is specialized in self-collected samples from previous studies. This procedure is considered feasible based on data showing that the dry brush is analytically stable for HPV DNA detection for up to 32 weeks at temperatures ranging from 4 ºC to 30 ºC. After HPV analyses, residual material from the self-collected samples will be stored in a biobank in Denmark at Aarhus University hospital and saved for future research.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive (women with HIV-1, HIV-2 AND HIV1/2 are all eligible)
* Age between 18 and 65 years

Exclusion Criteria:

* Current pregnancy
* Pregnancy within the last 3 months
* Prior hysterectomy
* Women using other vaginal products than contraceptives and water based lubricants
* Women who don't understand the extent of the study
* Bleeding due to ongoing period

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study is part of an international collaboration between the Department of Infectious Medicine at Aarhus University Hospital, the Bandim Health Project in Guinea-Bissau and Belgian researchers. Bandim Health project is a health and demographic surveillance system site that follows a population of more than 200.000 individuals in Guinea-Bissau. That population has created the base for the Guinea-Bissau Nationwide HIV-cohort with more than 35.000 patients.
  The patients are provided free HIV-treatment and follow-up in the country. There is currently 9 large HIV-clinics in the country, and women presenting at these clinics will be invited to enroll if they meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 502 (Actual)
Dates: Start 2023-05-29 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of implementing HPV self sampling for cervical cancer screening | April 2023 - February 2024
  Among women meeting the inclusion criteria, the investigators want to estimate the prevalence of how many accepts the offer to collect self-samples, thereby gaining knowledge on the feasibility of implementing self-sampling as a cervical cancer screening method in Guinea-Bissau.
HPV-prevalence among HIV-infected women in Guinea-Bissau | April 2023 - February 2024
  The investigators want to estimate the prevalence of high risk HPV infection among HIV-infected women in the Nationwide HIV-cohort in Guinea-Bissau.

SECONDARY OUTCOMES:
Experiences with self-collected vaginal and urine samples | April 2023 - February 2024
  Among the women accepting the invitation to enroll in the study, the investigators will through a questionnaire obtain data on the participants experiences with the two self-sampling devices.
HPV-genotype agreement between vaginal- and urine samples | April 2023 - February 2024
  Among HPV-positive women the investigators want to describe the genotype agreement among the two sample types

CONTACTS AND LOCATIONS:
Overall Officials: Sanne Jespersen, MD, PhD, Principal Investigator — Department of infectious diseases, Aarhus University Hospital, Denmark
Locations (1):
- Centro Tratamento Ambúlatorios na Guinea-Bissau, Bissau, Guinea-Bissau

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Background] Chaturvedi AK, Madeleine MM, Biggar RJ, Engels EA. Risk of human papillomavirus-associated cancers among persons with AIDS. J Natl Cancer Inst. 2009 Aug 19;101(16):1120-30. doi: 10.1093/jnci/djp205. Epub 2009 Jul 31. PMID 19648510
- [Background] Hawes SE, Critchlow CW, Faye Niang MA, Diouf MB, Diop A, Toure P, Aziz Kasse A, Dembele B, Salif Sow P, Coll-Seck AM, Kuypers JM, Kiviat NB. Increased risk of high-grade cervical squamous intraepithelial lesions and invasive cervical cancer among African women with human immunodeficiency virus type 1 and 2 infections. J Infect Dis. 2003 Aug 15;188(4):555-63. doi: 10.1086/376996. Epub 2003 Jul 23. PMID 12898443
- [Background] Mezei AK, Armstrong HL, Pedersen HN, Campos NG, Mitchell SM, Sekikubo M, Byamugisha JK, Kim JJ, Bryan S, Ogilvie GS. Cost-effectiveness of cervical cancer screening methods in low- and middle-income countries: A systematic review. Int J Cancer. 2017 Aug 1;141(3):437-446. doi: 10.1002/ijc.30695. Epub 2017 Apr 3. PMID 28297074
- [Background] Wright TC, Stoler MH, Behrens CM, Sharma A, Zhang G, Wright TL. Primary cervical cancer screening with human papillomavirus: end of study results from the ATHENA study using HPV as the first-line screening test. Gynecol Oncol. 2015 Feb;136(2):189-97. doi: 10.1016/j.ygyno.2014.11.076. Epub 2015 Jan 8. PMID 25579108
- [Background] Gilham C, Sargent A, Kitchener HC, Peto J. HPV testing compared with routine cytology in cervical screening: long-term follow-up of ARTISTIC RCT. Health Technol Assess. 2019 Jun;23(28):1-44. doi: 10.3310/hta23280. PMID 31219027
- [Background] Coorevits L, Traen A, Binge L, Van Dorpe J, Praet M, Boelens J, Padalko E. Are vaginal swabs comparable to cervical smears for human papillomavirus DNA testing? J Gynecol Oncol. 2018 Jan;29(1):e8. doi: 10.3802/jgo.2018.29.e8. PMID 29185266
- [Background] Boggan JC, Walmer DK, Henderson G, Chakhtoura N, McCarthy SH, Beauvais HJ, Smith JS. Vaginal Self-Sampling for Human Papillomavirus Infection as a Primary Cervical Cancer Screening Tool in a Haitian Population. Sex Transm Dis. 2015 Nov;42(11):655-9. doi: 10.1097/OLQ.0000000000000345. PMID 26462192
- [Background] Jun JK, Lim MC, Hwang SH, Shin HY, Hwang NR, Kim YJ, Yoo CW, Lee DO, Joo J, Park SY, Lee DH. Comparison of DRY and WET vaginal swabs with cervical specimens in Roche Cobas 4800 HPV and Abbott RealTime High Risk HPV tests. J Clin Virol. 2016 Jun;79:80-84. doi: 10.1016/j.jcv.2016.04.012. Epub 2016 Apr 23. PMID 27111579
- [Background] Van Keer S, Latsuzbaia A, Vanden Broeck D, De Sutter P, Donders G, Doyen J, Tjalma WAA, Weyers S, Arbyn M, Vorsters A. Analytical and clinical performance of extended HPV genotyping with BD Onclarity HPV Assay in home-collected first-void urine: A diagnostic test accuracy study. J Clin Virol. 2022 Oct;155:105271. doi: 10.1016/j.jcv.2022.105271. Epub 2022 Aug 24. PMID 36049283
- [Background] Tranberg M, Jensen JS, Bech BH, Andersen B. Urine collection in cervical cancer screening - analytical comparison of two HPV DNA assays. BMC Infect Dis. 2020 Dec 4;20(1):926. doi: 10.1186/s12879-020-05663-7. PMID 33276740
- [Background] Tranberg M, Bech BH, Blaakaer J, Jensen JS, Svanholm H, Andersen B. Preventing cervical cancer using HPV self-sampling: direct mailing of test-kits increases screening participation more than timely opt-in procedures - a randomized controlled trial. BMC Cancer. 2018 Mar 9;18(1):273. doi: 10.1186/s12885-018-4165-4. PMID 29523108
- [Background] Tranberg M, Jensen JS, Bech BH, Blaakaer J, Svanholm H, Andersen B. Good concordance of HPV detection between cervico-vaginal self-samples and general practitioner-collected samples using the Cobas 4800 HPV DNA test. BMC Infect Dis. 2018 Jul 27;18(1):348. doi: 10.1186/s12879-018-3254-y. PMID 30053836
- [Derived] Madsen KL, Tranberg M, Norgaard P, Medina C, Storgaard M, Vorsters A, Van Keer S, Honge BL, Jespersen S. Feasibility of First-Void Urinary and Vaginal Self-Sampling for High-Risk Human Papillomavirus Testing Among Women Living With Human Immunodeficiency Virus in Guinea-Bissau-A Multicenter Cross-Sectional Study. J Med Virol. 2025 Jul;97(7):e70466. doi: 10.1002/jmv.70466. PMID 40590686
- See also: WHO Cervical Cancer elimination Strategy — https://www.who.int/initiatives/cervical-cancer-elimination-initiative